CLINICAL TRIAL: NCT07013461
Title: International Collaborative Study to Develop the AJCC/UICC TNM Version-Ten for Nasopharyngeal Cancer
Brief Title: International Collaborative Study on AJCC/UICC TNM-10 for Nasopharyngeal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: The University of Hong Kong-Shenzhen Hospital (Other)
Collaborators: Sun Yat-sen University Cancer Hosptial (Unknown); Fujian Cancer Hospital (Other Government); Chinese Academy of Medical Sciences (Other); Jiangxi Provincial Cancer Hospital (Other); Zhejiang Cancer Hospital (Other); Chongqing University Cancer Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Sichuan Cancer Hospital and Research Institute (Other); First Affiliated Hospital of Fujian Medical University (Other); Queen Mary Hospital, Hong Kong (Other); The Queen Elizabeth Hospital (Other); Pamela Youde Nethersole Eastern Hospital (Other); Tuen Mun Hospital, Hospital Authority, Hong Koong (Unknown); Princess Margaret Hospital, Hong Kong (Other Government); United Christian Hospital (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Anne Wing-mui Lee, Consultant, Clinical Cancer Center, The University of Hong Kong-Shenzhen Hospital
Other Study IDs: hkuszh2025075
Record Dates: First submitted 2025-06-01; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Nasopharyngeal Cancinoma (NPC)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with histologically confirmed NPC: All enrolled patients will receive diagnosis and treatment according to the standard clinical practice of each participating center.

SUMMARY:
The goal of this international, multicenter, prospective observational study is to improve prognostication and prediction of failure pattern for nasopharyngeal carcinoma (NPC), in order to provide more accurate guidance for personalized treatment decision. Firstly, we aim to improve the fundamental TNM staging system (current AJCC/UICC TNM Version-Nine) based on universally assessable anatomical parameters. Secondly, we aim to further refine prognostication for individual patients by integrating anatomical TNM parameters with non-anatomical factors and molecular biomarkers. In addition to the core group of participating centers from China (including Hong Kong) where NPC is most prevalent, the study will enrol patients from multiple countries/regions including those from non-endemic areas to provide global data. Patients treated with contemplary treatment methods during October 2025 to September 2026 will be recruited and they will be followed up for 5 years to generate detailed records for robust evaluation.

Key Questions:

* To achieve optimal improvement of anatomically based AJCC/UICC TNM Classification for global application
* To achieve precise prediction of failure pattern for individual patients by integration of TNM system and non-anatomical prognostic factors/molecular biomarkers Recruited patients with confirmed histological diagnosis of NPC will undergo standard clinical evaluations and receive treatment per institutional guidelines.

The anatomical extent of disease at presentation will be evaluated by experienced radiologists and oncologists. The patient will be followed up for 5 years and clinical outcome will be recorded for analyses on correlation with prognostic factors.

This study will be another important milestone for NPC staging because firstly, this is the first time that the data are based on prospective data to ensure comprehensive coverage of all essential evidence; and secondly, this is the first time that centers from non-endemic countries/regions will also participate to ensure that the final recommendations are globally applicable. The findings will provide valuable evidence for the development of the AJCC/UICC TNM Version-Ten staging system and prognostic system to improve risk stratification for designing personalized treatment strategy, ultimately leading to improvement of patient outcome and patient selection for future research worldwide.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is an Epstein-Barr virus-associated malignancy with a striking geographical predominance, over 70% of global cases occur in East and Southeast Asia. The current AJCC/UICC TNM Version-Nine staging system, launched in January 2025, is a significant advancement in prognostic stratification. The recommendations are based by high quality retrospective data from Mainland China and Hong Kong and consensus building among international multidisciplinary experts, taking into consideration both the statistical evidence of benefit and clinical applicability.

Recent years have witnessed transformative changes in NPC treatment paradigms, including advancements in radiotherapy techniques, the integration of immune checkpoint inhibitors, and intensified treatment for metastatic disease. In addition, studies have demonstrated the independent prognostic value of non-anatomical factors such as circulating EBV DNA levels, and various hematologic biomarkers. These developments necessitate continual improvement of the TNM staging system to align with contemporary management with diagnostic and therapeutic advancements.

This international, multicenter, prospective observational study is designed to address these critical requirements to generate high-quality evidence for developing the next generation TNM staging system (AJCC/UICC Version-Ten). The study will enroll all consecutive histopathological confirmed NPC patients treated during October 2025 and September 2026 from leading cancer centers worldwide. Detailed data on clinicopathological characteristics, imaging findings, molecular markers (including EBV-DNA), treatment and outcome will be collected and analyzed.

The primary endpoint of the study is overall survival (OS), while secondary endpoints focus on the pattern of failure at different sites: local failure-free survival (L-FFS), regional nodal failure-free survival (N-FFS), and distant failure-free survival (D-FFS). Correlation of these outcomes to anatomical and non-anatomical factors will be analyzed.

This study will be another important milestone for NPC staging because firstly, this is the first time that the data are based on prospective data to ensure comprehensive coverage of all essential evidence; and secondly, this is the first time that centers from non-endemic countries/regions will also participate to ensure that the final recommendations are globally applicable. The findings will provide valuable evidence for the development of the AJCC/UICC TNM Version-Ten staging system and prognostic system to improve risk stratification for designing personalized treatment strategy, ultimately leading to improvement of patient outcome and patient selection for future research worldwide.

ELIGIBILITY:
Inclusion Criteria:

* All histologically confirmed nasopharyngeal carcinoma treated between 1 Oct 2025 and 30 Sep 2026

Exclusion Criteria:

* Non-epithelial tumors of nasopharynx (including lymphoma, sarcoma of soft tissue, bone/cartilagetumors. mucosal melanoma, salivary type tumors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in participating centers
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  The time to death for any cause

SECONDARY OUTCOMES:
Local Failure Free Survival (LFFS) | 5 years
  The time to local tumor persistence/recurrence.
Regional Nodal Failure Free Survival (N-FFS) | 5 years
  The time to regional nodal persistence/recurrence
Distant Failure-Free Survival (D-FFS) | 5 years
  The time to the first occurrence of distant metastases